CLINICAL TRIAL: NCT02237716
Title: Rapid Intravenous Infusion of Mannitol Results in a Dipper-type Change in Stroke Volume Variation in Patients Undergoing Major Neurosurgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xinxin Shao, Resident, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: MN2014
Record Dates: First submitted 2014-08-26; First posted 2014-09-11 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Craniotomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to observe the variation of Hemodynamics、lactic acid、base excess、peripheral vascular resistance and DO2 through FloTrac™/Vigileo™ system after rapid infusion mannitol in neurosurgery.The hemodynamic changes after mannitol infusion are shown in Figure 1. HR (Fig. 1A) and systolic BP (Figure 1B) significantly increased between 0 min and 10 min (P = 0.041) and between -10 min and 10 min (P = 0.073), respectively; these two variables decreased steadily and returned to the baseline. Diastolic BP (Fig. 1B) showed no significant change after mannitol infusion (P = 0.102). CVP (Fig. 1C) significantly increased between -20 min and 0 min (P < 0.001) and constantly decreased after 0 min, which remained below the baseline between 30 min and 60 min. CI (Fig. 1D) and SVI (Fig. 1E) showed a significant persistent increase between -20 min to 0 min (P < 0.001) and between -20 min and 10 min (P < 0.001), respectively. SVV exhibited a dipper-type change shown as a significant decrease between -20 min and 0 min and a significant increase between 0 min and 60 min (P < 0.001), which returned to the baseline after 20 min.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria were: being aged between 16 and 70 years;
* with a body mass index of 18-25 kg/m2;
* with a physical status classified as ASA class I or II;
* and scheduled for elective craniotomy

Exclusion Criteria:

* Any patient would be excluded from this study if the patient had complicating serious coagulopathy, hepatorenal insufficiency, aortic regurgitation, or cardiac arrhythmia;
* had a previous history of intra-aortic balloon counterpulsation;
* exhibited systolic blood pressure (SBP) ≥160 mmHg, diastolic blood pressure (DBP) ≥100 mmHg, or heart rate ≥ 100 bpm on operating room admission;
* or rejected to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: scheduled for elective craniotomy
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2014-06; Primary Completion 2014-12 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
cardiac index | during the procedure
stroke volume index | during the procedure
stroke volume variation | during the procedure
systolic pressure | during the procedure
central venous pressure | during the procedure
heart rate | during the procedure
peripheral vascular resistance | during the procedure

SECONDARY OUTCOMES:
base excess | during the procedure
lactic acid | during the procedure
DO2I | during the procedure